CLINICAL TRIAL: NCT00761436
Title: Stereotactic Intrastriatal Implantation of Spheramine in Advanced Parkinson's Disease Patients: A Pilot Study of Tolerability and Efficacy.
Brief Title: Pilot Study of Safety and Efficacy of Spheramine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was completed, only life long extended follow-up phase was discontinued after 12 years
Sponsor: Bayer (Industry)
Collaborators: Titan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91677; 311361 (Other: Company Internal)
Record Dates: First submitted 2008-09-26; First posted 2008-09-29 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Parkinson''s Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Biological: Spheramine (BAY86-5280)

INTERVENTIONS:
Biological: Spheramine (BAY86-5280) — Stereotactic Intrastriatal Implantation

SUMMARY:
Tolerability and Efficacy of Spheramine will be evaluated after operative implantation (Stereotactic Intrastriatal Implantation) in patients with advanced Parkinson's Disease

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease (PD). As defined by:

  * presence of bradykinesia and either rest tremor or rigidity
  * history of asymmetry of PD signs
  * history of progression of PD signs, and
  * no other suspected cause of PD signs
* Patient is between 40 and 70 years of age, inclusive
* Patient is L-dopa-sensitive and has unequivocal clinical "off" periods as documented by home diary, completed on 4 consecutive days with an average of 1.5 hours/day in the clinically "off" state
* Patient is Hoehn & Yahr stage III or higher in the practically defined "off" phase
* All other medical problems are stable or under control and are not contraindications to general anesthesia or stereotactic neurosurgery
* Patient's brain magnetic imaging resonance (MRI) shows no abnormality that would contraindicate Spheramine implantation
* Patient does not have a major psychiatric problem or dementia
* Patient must give written informed consent to participate in this study
* Patient must be on a stable dose of antiparkinsonian medication for at least 1 month prior to completion of the home diary assessment and the baseline UPDRS assessments
* If the patient is a woman of childbearing potential, she must not be nursing or pregnant and must use an adequate form of birth control for the duration of the study deemed appropriate by the investigator such as oral contraceptives, IUD, or condoms
* Patient must be living with or in close constant contact with a person who can contribute information as to the patient's condition before and after implant and provide assistance, if necessary

Exclusion Criteria:

* Patients with atypical Parkinson's disease (e.g. parkinsonian "plus" syndrome, secondary Parkinsonian syndrome)
* Patients exhibiting only a tremor-based symptomatology
* Patients exhibiting very severe dyskinesias (lasting more than 2 hour/day) exacerbated by L-dopa, evaluated as 4/4 on the dyskinesia scale (violent dyskinesias, incompatible with any normal motor task)
* Women of childbearing potential without contraception
* Patients who are non-cooperative or incapable of completing self-evaluation scales or diaries
* Patients presenting with known pharmacologic immunosuppression related to chemotherapeutic treatment for malignancy, autoimmune disease, allografts or other medical conditions associated with immunosuppression
* Patient's cardiovascular, pulmonary, renal and hematological state contraindicates use of general anesthesia
* Evidence of abnormal coagulation including PT > 13 sec, PT > 35 sec or platelets < 5 ml
* Patients having had previous stereotactic brain surgery
* Patients treated by apomorphine pump
* Patients with significant cognitive impairment, untreated or treatment resistant depression, psychosis, hallucinations or delusions that would prevent their effective participation in the study
* Patients who have participated in another experimental drug or device trial in the past 30 days

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2000-02-29 (Actual); Primary Completion 2012-05-14 (Actual); Study Completion 2012-05-14 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for evaluating efficacy will be the motor subscore of the Unified Parkinson's Disease Rating Scale (UPDRS) (version 3.0) in the practically defined "off" state. During the Screening and at Baseline Evaluations. | Evaluations, and at approximately 1, 3, 6, 9, 12, 15, 18 and 24 months post-implantation and annually thereafter, the patients Parkinson's symptomatology will be evaluated both on their baseline drug therapy and in the practically defined "off" period.

SECONDARY OUTCOMES:
Involuntary Movements, time Motor Tests | Performed during defined "off" and best "on" states
Motor Fluctuation and Percent OFF Time Evaluation | Daily "on" phases, "off" phases and hours of sleep per day, using Home Diary
Quality of Life and Physician's and Patients Global Evaluations | Every visit until year 5
Neuropsychological Evaluations | Will occur pre-operatively and at 3, 12 and 24 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Atlanta, Georgia, United States